CLINICAL TRIAL: NCT05092828
Title: Does Intrathecal Morphine Affect Outcomes in Spine Deformity Surgery: A Prospective, Randomized Clinical Controlled Trial
Brief Title: Does Intrathecal Morphine Affect Outcomes in Spine Deformity Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sonoran Spine Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Michael Chang, MD, Clinical Associate Professor, Sonoran Spine Research and Education Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SS-MSC-001
Record Dates: First submitted 2021-09-16; First posted 2021-10-26 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Analgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Nursing staff and physical therapists will be blinded to intrathecal morphine utilization as to not bias the input of these variables
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): Patients in this group will receive intrathecal morphine in addition to standard post-operative pain medications
  Interventions: Drug: Intrathecal Morphine Injection
- Control Group (Active Comparator): Patients in this group will receive standard post-operative pain medications but will not receive intrathecal morphine
  Interventions: Drug: Pain Relieving

INTERVENTIONS:
Drug: Intrathecal Morphine Injection — In addition to standard post-operative pain management, Intratechal morphine will be given to patients in this group.
  Other Names: Subarachnoid injection of morphine
  Arms: Study Group
Drug: Pain Relieving — Patient in this group will receive standard postoperative pain medications other than inthrathecal injection of morphine
  Other Names: Standard Post-operative pain medications other than intrathecal morphine
  Arms: Control Group

SUMMARY:
This study aims to compare the effects of intrathecal morphine to traditional pain management strategies on post-operative recovery for deformity surgery.

DETAILED DESCRIPTION:
Background Deformity surgery is considered one of the most painful procedures patients can undergo in medicine today. Stringent protocols for pain management have done much to dramatically increase patient satisfaction, but the procedure still lags considerably behind advances in pain control when compared to other procedures such as total joint surgery. Specifically, it has been reported that over half of patients undergoing spine surgery report inadequate pain control the first 24 hours after surgery. Uncontrolled pain has been shown to correlate with prolonged hospital stays, delayed ambulation, poor functional outcomes, and increased risk for the development of chronic pain. Furthermore, the large amount of narcotics given to patients in an attempt to mitigate their pain postoperatively often leads to significant complications in their own right, such as ileus, mental status changes, and nausea. New modalities to treat postoperative pain, especially in the initial days following deformity correction, are needed.

Intrathecal (subarachnoid) injection of morphine has been used to treat severe pain since the 1970's. Its efficacy in treating postoperative pain has been well documented in various specialties including obstetrics, oncology, general surgery, and orthopedic surgery. Specific to spine surgery, intrathecal morphine is an attractive option given the access and visualization of the thecal sac in addition to the high demand of pain control required postoperatively. However, there remains no definitive consensus regarding the use of intrathecal morphine in spine surgery. Current literature is limited by few randomized trials, small sample sizes, heterogeneity of outcomes recorded, and an unclear association with complications. Additionally, there is a paucity of data dedicated to patients undergoing deformity correction. Accordingly, there is a need for high-quality trials to investigate the role of intrathecal morphine in adult spinal deformity surgery.

In this study, we hypothesized that the use of intrathecal morphine will significantly reduce post-operative pain after deformity surgery, reduce opioid utilization, decrease hospital stay, allow for earlier ambulation, increase patient satisfaction, and have comparable complications to traditional pain management strategies. This study aims to compare the effects of intrathecal morphine to traditional pain management strategies on post-operative recovery for deformity surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years and older with a diagnosis of adult or degenerative scoliosis,
* Patients meeting criteria for surgical correction involving back and/or leg pain
* Fusion of 4+ levels,
* Competency to undergo informed consent process,
* Medical clearance for spinal fusion surgery,

Exclusion Criteria:

* Patients with lumbar spine inaccessible for intrathecal Duragesic (fused L2-S1)
* Patients undergoing 3 or less levels of fusion
* Patients with neuromuscular disease
* Opioid intolerance or dependence
* Severe coexisting diseases
* ASA III

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-02 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Pain and Outcome Assessment | preoperative
  postoperative pain using Numerical pain score 0 no pain - 10 severe intolerable pain Oswesty Disability Index and Scoliosis Research Society Questionnaire
Pain and Outcome Assessment | 6 week, post operative
  postoperative pain using Numerical pain score 0 no pain - 10 severe intolerable pain
Pain and Outcome Assessment | 3 months post operative
  postoperative pain using Numerical pain score 0 no pain - 10 severe intolerable pain
Pain and Outcome Assessment | 1 year post operative
  postoperative pain using Numerical pain score 0 no pain - 10 severe intolerable pain
Pain and Outcome Assessment | 2-year follow up
  postoperative pain using Numerical pain score 0 no pain - 10 severe intolerable pain

SECONDARY OUTCOMES:
Pain medications | Preoperative
  Types of pain medication (Narcotics or Non-Narcotics)
Pain medications | 6 weeks Post Operative
  Types of pain medication (Narcotics or Non-Narcotics)
Pain medications | 3 months Post Operative
  Types of pain medication (Narcotics or Non-Narcotics)
Pain medications | 1 year Post Operative
  Types of pain medication (Narcotics or Non-Narcotics)
Pain medications | 2 year Post Operative
  Types of pain medication (Narcotics or Non-Narcotics)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Chang, MD, Principal Investigator — Sonoran Spine Research and Education Foundation; Andrew Chung, DO, Principal Investigator — Sonoran Spine Research and Education Foundation
Locations (2):
- United States (2):
  - Sonoran Spine in Collaboration with HonorHealth, Tempe, Arizona
  - Sonoran Spine, Tempe, Arizona